CLINICAL TRIAL: NCT01549067
Title: The Real Clinical Background of Advanced Colorectal Cancer Treatment Situation Survey
Acronym: Sprit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Medical Doctor Association (Other)
Responsible Party: Principal Investigator, Lin Shen，MD & Ruihua Xu，MD、PhD, Principal Investigator, Chinese Medical Doctor Association
Other Study IDs: Sprit
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Malignant Neoplasm; Colorectal Cancer
Keywords: Advanced; Colorectal Cancer; Targeted chemotherapy; Surgery; Radiotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Collect the real clinical background of advanced colorectal cancer c of China.

DETAILED DESCRIPTION:
The Primary Objectives of this study is collect the real clinical background of advanced colorectal cancer treatment situation of China. The Secondary Objectives is the mutation of K-ras , targeting therapy , use present situation of cetuximab and liver metastases treatment situation of colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of metastatic colorectal cancer.

Exclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis other than metastatic colorectal cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Advanced Colorectal Cancer
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Zhongshan, Guangzhou